CLINICAL TRIAL: NCT00005999
Title: A Phase II Study of Arsenic Trioxide (NSC #706363) in Patients With Advanced Cervical Carcinoma
Brief Title: Arsenic Trioxide in Treating Patients With Stage IVB or Recurrent Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068003; MSKCC-00018; NCI-30
Record Dates: First submitted 2000-07-05; First posted 2003-05-21 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2002-03

CONDITIONS: Cervical Cancer
Keywords: recurrent cervical cancer; stage IVB cervical cancer; cervical squamous cell carcinoma; cervical adenocarcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Arsenic Trioxide

INTERVENTIONS:
Drug: arsenic trioxide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of arsenic trioxide in treating patients who have stage IVB or recurrent cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the efficacy of arsenic trioxide in patients with stage IVB or recurrent cervical carcinoma.
* Determine the safety of this treatment in these patients.

OUTLINE: Patients receive arsenic trioxide IV over 1-4 hours on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 12-37 patients will be accrued for this study over 10-19 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IVB or recurrent cervical carcinoma that is not amenable to standard curative therapies

  * Squamous carcinoma OR
  * Adenocarcinoma
* Measurable disease

  * At least 20 mm by conventional techniques OR
  * At least 10 mm by spiral CT scan
  * Nonmeasurable disease defined as any of the following:

    * Bone disease
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Inflammatory breast disease
    * Lymphangitis cutis/pulmonis
    * Abdominal masses not confirmed or followed by imaging techniques
    * Cystic lesions
* No active brain metastases

PATIENT CHARACTERISTICS:

Age:

* 17 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Greater than 3 months

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST and ALT no greater than 2.5 times ULN

Renal:

* Creatinine no greater than 2.0 mg/dL OR
* Creatinine clearance at least 50 mL/min

Cardiovascular:

* No cardiac arrhythmias, unstable angina, or conduction abnormalities
* No New York Heart Association class III or IV heart disease or clinical evidence of congestive heart failure
* Pretreatment QTc less than 500 msec

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 4 months after study
* No grade 3 or greater neurologic abnormalities
* No history of seizures
* No concurrent uncontrolled active infection

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No more than 2 prior therapies for advanced disease

Chemotherapy:

* No more than 2 prior therapies for advanced disease
* At least 4 weeks since prior chemotherapy

Endocrine therapy:

* No more than 2 prior therapies for advanced disease

Radiotherapy:

* No more than 2 prior therapies for advanced disease
* At least 4 weeks since prior radiotherapy

Surgery:

* Not specified

Other:

* At least 4 weeks since prior cytotoxic therapy or investigational agents

Min Age: 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-04; Study Completion 2003-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol Aghajanian, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States